CLINICAL TRIAL: NCT03430843
Title: A Randomized, Controlled, Open-label, Global Phase 3 Study Comparing the Efficacy of the Anti-PD-1 Antibody Tislelizumab (BGB-A317) Versus Chemotherapy as Second Line Treatment in Patients With Advanced Unresectable/Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: A Study of Tislelizumab (BGB-A317) Versus Chemotherapy as Second Line Treatment in Participants With Advanced Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-302; 2017-003699-30 (EudraCT Number); CTR20171026 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2018-01-29; First posted 2018-02-13 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: Unresectable; metastatic; second-line; squamous; esophagus; chemotherapy; paclitaxel; docetaxel; irinotecan
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Neoplasm Metastasis | interventions — tislelizumab; Paclitaxel; Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tislelizumab (Experimental): Tislelizumab on Day 1, given every 21 days
  Interventions: Drug: Tislelizumab
- Investigator chosen chemotherapy (ICC) (Active Comparator): Paclitaxel on Day 1, given every 21 days or on a weekly schedule; OR Docetaxel on Day 1, given every 21 days; OR Irinotecan on Days 1 and 8, given every 21 days
  Interventions: Drug: Paclitaxel; Drug: Docetaxel; Drug: Irinotecan

INTERVENTIONS:
Drug: Tislelizumab — 200 mg administered intravenously (IV)
  Other Names: BGB-A317
  Arms: Tislelizumab
Drug: Paclitaxel — 135-175 mg /m² administered IV , or 80-100 mg/m^2 administered IV according to local guidelines for standard of care
  Arms: Investigator chosen chemotherapy (ICC)
Drug: Docetaxel — 75 mg/m^2 administered IV or 70 mg/m^2 IV in Japan
  Arms: Investigator chosen chemotherapy (ICC)
Drug: Irinotecan — 125 mg/m^2 administered IV
  Arms: Investigator chosen chemotherapy (ICC)

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of tislelizumab as second line treatment in participants with advanced unresectable/metastatic ESCC that had progressed during or after first line therapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed diagnosis of esophageal squamous cell carcinoma (ESCC)
2. Tumor progression during or after first-line treatment for advanced unresectable / metastatic ESCC
3. At least one measurable/evaluable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 prior to randomization

Key Exclusion Criteria:

1. Receipt of 2 or more prior systemic treatments for advanced/metastatic unresectable ESCC
2. History of gastrointestinal perforation and /or fistula or aorto-esophageal fistula within 6 months prior to randomization
3. Tumor invasion into organs located adjacent to the esophageal disease site (eg, aorta or respiratory tract) at an increased risk of fistula in the study treatment assessed by investigator
4. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage
5. Received prior therapies targeting programmed death 1 (PD-1) or programmed death ligand 1 (PD-L1)
6. Prior malignancy active within the previous 2 years (exceptions include the tumor under investigation in this trial, and locally recurring cancers that have undergone curative treatment, such as resected basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the prostate, cervix or breast)
7. Active brain or leptomeningeal metastasis.
8. Has active autoimmune disease or history of autoimmune diseases at high risk for relapse
9. Known history of, or any evidence of interstitial lung disease, non-infectious pneumonitis, pulmonary fibrosis diagnosed based on imaging or clinical findings, or uncontrolled systemic diseases, including diabetes, hypertension, acute lung diseases, etc
10. Known history of Human Immunodeficiency Virus (HIV)
11. Has cardiovascular risk factors
12. Pregnant or breastfeeding woman.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (104):
- United States (2):
  - Henry Ford Hospital, Detroit, Michigan
  - Toledo Clinic Cancer Center, Toledo, Ohio
- Belgium (4):
  - Imelda Ziekenhuis Bonheiden, Bonheiden
  - Cliniques Universitaires Saint Luc, Brussels
  - Uz Antwerpen, Edegem
  - University Hospitals Leuven, Leuven
- China (38):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - Huaian Second Peoples Hospital, Huaian, Jiangsu
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital Branch South, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiangxi Province Cancer Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Provincial Peoples Hospital, Taiyuan, Shanxi
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- France (10):
  - Chru de Brest Hospital Morvan, Brest
  - Centre Georges Francois Leclerc, Dijon
  - Chu Besancon Hopital Jean Minjoz, Doubs
  - Centre Oscar Lambret, Lille
  - Hopital Prive Jean Mermoz, Lyon
  - Icm Val Daurelle, Montpellier
  - Chu Bordeaux Hopital Haut Leveque, Pessac
  - Chu de Poitiers Site de La Mileterie, Poitiers
  - Ico Site Rene Gauducheau, SaintHerblain
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Charite Universitatsmedizin Berlin, Berlin
  - Universitares Krebszentrum Leipzig, Leipzig
  - Klinikum Johannes Gutenberg Universitaet Mainz, Mainz
- Italy (5):
  - Ospedale Di Faenza, Faenza
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori Irst, Meldola
  - Azienda Ospedaliero Universitaria San Luigi Gonzaga, Orbassano
  - Aou Pisana, Stabilimento Di Santa Chiara, Pisa
  - Ao Citta Della Salute E Della Scienza Di Torino Presidio O, Torino
- Japan (17):
  - Akita University Hospital, Akitashi, Akita
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Nho Shikoku Cancer Center, Matsuyama, Ehime
  - Nho Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - St Marianna University School of Medicine Hospital, Yokohama, Kanagawa
  - Osaka International Cancer Institute, Osakashi, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suitashi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsukishi, Osaka
  - Saitama Cancer Center, Kitaadachigun, Saitama
  - Shizuoka Cancer Center, Suntogun, Shizuoka
  - National Cancer Center Hospital, Chuoku, Tokyo
  - Cancer Institute Hospital of Jfcr, Kotoku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Kochi Health Sciences Center, Kochi
  - Kyoto University Hospital, Kyoto
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Incheon Gwang'yeogsi
  - Chonnam National University Hwasun Hospital, HwasunGun, Jeollanam-do
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - Korea University Guro Hospital, Seoul, Seoul Teugbyeolsi
- Spain (8):
  - Hospital Del Mar, Barcelona
  - Hospital Universitario Vall Dhebron, Barcelona
  - Institut Catala Doncologia, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario de Octubre, Madrid
  - Hospital Universitario Hm Madrid Sanchinarro, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi Mei Hospital Liouying, Tainan
  - National Taiwan University Hospital East Campus, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (6):
  - The Christie Hospital, Greater Manchester
  - Guys and St Thomas Hospital Nhs Foundation Trust, London
  - Sarah Cannon Research Institute Uk, London
  - St Marys Hospital Imperial College Healthcare Nhs Trust, London
  - Mount Vernon Hospital (Mount Vernon Cancer Center), Northwood
  - Royal Marsden Nhs Foundation Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Shen L, Kato K, Kim SB, Ajani JA, Zhao K, He Z, Yu X, Shu Y, Luo Q, Wang J, Chen Z, Niu Z, Zhang L, Yi T, Sun JM, Chen J, Yu G, Lin CY, Hara H, Bi Q, Satoh T, Pazo-Cid R, Arkenau HT, Borg C, Lordick F, Li L, Ding N, Tao A, Shi J, Van Cutsem E; RATIONALE-302 Investigators. Tislelizumab Versus Chemotherapy as Second-Line Treatment for Advanced or Metastatic Esophageal Squamous Cell Carcinoma (RATIONALE-302): A Randomized Phase III Study. J Clin Oncol. 2022 Sep 10;40(26):3065-3076. doi: 10.1200/JCO.21.01926. Epub 2022 Apr 20. PMID 35442766
- [Derived] Ajani JA, Wang K, Nikolaidis GF, Coaquira Castro J, Augusto Novis de Figueiredo M, Sun JM, Soulanis K, Tasoulas A, Zhan L. Comparative Efficacy and Safety of Tislelizumab in Second-Line Esophageal Squamous Cell Carcinoma: Systematic Literature Review and Simulated Treatment Comparisons. Adv Ther. 2025 Dec 3. doi: 10.1007/s12325-025-03410-5. Online ahead of print. PMID 41335329
- [Derived] Lu Z, Du W, Jiao X, Wang Y, Shi J, Shi Y, Shu Y, Niu Z, Hara H, Wu J, Hsu CH, Van Cutsem E, Brock MV, Zhang Z, Ding N, Zhang Y, Shen Z, Shen L. NOTCH1 Mutation and Survival Analysis of Tislelizumab in Advanced or Metastatic Esophageal Squamous Cell Carcinoma: A Biomarker Analysis From the Randomized, Phase III, RATIONALE-302 Trial. J Clin Oncol. 2025 Jun;43(16):1898-1909. doi: 10.1200/JCO-24-01818. Epub 2025 Apr 3. PMID 40179324
- [Derived] He Q, Shi X, Yan J, Wu M, Gu C, Yu X. Circulating tumor DNA serial monitoring of relapse and responses to tislelizumab immunotherapy as second-line monotherapy for metastatic esophageal squamous cell carcinoma: A prospective study. Mol Clin Oncol. 2024 Feb 9;20(4):29. doi: 10.3892/mco.2024.2727. eCollection 2024 Apr. PMID 38414510
- [Derived] Hara H, Satoh T, Kojima T, Tsushima T, Sunakawa Y, Okada M, Ding N, Wu H, Li L, Yu T, Barnes G, Kato K. Second-line tislelizumab versus chemotherapy in Japanese patients with advanced or metastatic esophageal squamous cell carcinoma: subgroup analysis from RATIONALE-302. Esophagus. 2024 Apr;21(2):102-110. doi: 10.1007/s10388-023-01040-w. Epub 2024 Jan 19. PMID 38240916
- [Derived] Kim SB, Van Cutsem E, Ajani J, Shen L, Barnes G, Ding N, Tao A, Xia T, Zhan L, Kato K. Tislelizumab in advanced/metastatic esophageal squamous cell carcinoma: health-related quality of life in Asian patients. Curr Med Res Opin. 2024 Jan;40(1):69-75. doi: 10.1080/03007995.2023.2270894. Epub 2024 Jan 3. PMID 37846080
- [Derived] Van Cutsem E, Kato K, Ajani J, Shen L, Xia T, Ding N, Zhan L, Barnes G, Kim SB. Tislelizumab versus chemotherapy as second-line treatment of advanced or metastatic esophageal squamous cell carcinoma (RATIONALE 302): impact on health-related quality of life. ESMO Open. 2022 Aug;7(4):100517. doi: 10.1016/j.esmoop.2022.100517. Epub 2022 Jul 1. PMID 35785595

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 132 study centers in Mainland China, Taiwan, United States, France, Italy, Germany, Spain, Japan, South Korea, Belgium and the United Kingdom.
Groups:
- Tislelizumab: Tislelizumab 200 mg intravenously (IV) on Day 1 every 21 days until disease progression, unacceptable toxicity, or other discontinuation criteria were met.
- Investigator Chosen Chemotherapy: Investigator choice of either paclitaxel 135-175 mg /m² on Day 1 IV every 21 days or 80-100 mg/m^2 on a weekly schedule; docetaxel 75 mg/m^2 IV on Day 1 every 21 days; or irinotecan 125 mg/m^2 IV on Days 1 and 8 every 21 days
Period: Overall Study
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Started | 256 | 256
Treated | 255 | 240
Completed | 0 | 0
Not Completed | 256 | 256
Not completed — Death | 233 | 233
Not completed — Sponsor Decision | 17 | 6
Not completed — Withdrawal by Subject | 5 | 14
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy | Total
Number analyzed (Participants) | 256 | 256 | 512
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (8.41) | 61.8 (8.02) | 61.8 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 41 | 80
  Male | 217 | 215 | 432
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 252 | 252 | 504
  Unknown or Not Reported | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 201 | 207 | 408
  Race: White or Caucasian | 53 | 44 | 97
  Race: Not Reported | 1 | 0 | 1
  Race: Unknown | 1 | 2 | 3
  Race: Black or African American | 0 | 2 | 2
  Race: Other | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status Score [Count of Participants; unit: Participants] — Measure Description: ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 | 66 | 61 | 127
    1 | 190 | 195 | 385
PD-L1 Expression Status [Count of Participants; unit: Participants] — Measure Description: Programmed death ligand 1 (PD-L1) positive is defined as visually-estimated Combined Positive Score (vCPS) >= 10%, PD-L1 negative is defined as vCPS < 10%, PD-L1 missing refers to the participants without sample collection, not evaluable at baseline, or scored with unqualified sample.
  Note terminology was updated from vCPS to Tumor Area Positivity (TAP) score in manuscripts.
  Participants
    vCPS >= 10% | 80 | 62 | 142
    vCPS < 10% | 100 | 122 | 222
    Missing | 76 | 72 | 148

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in the Intent-to-Treat (ITT) Analysis Set
Description: OS is defined as the length of time from the date of randomization until the date of death due to any cause in all randomized participants
Time Frame: Approximately 2 years and 10 months from date of first randomization
Population: The ITT analysis set included all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 256 | 256
Months | 8.6 [7.5 to 10.4] | 6.3 [5.3 to 7.0]
Statistical Analysis 1: Comparison: Tislelizumab vs Investigator Chosen Chemotherapy; Test type: Superiority; p = 0.0001, 1-sided, Log Rank Test; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.57 to 0.85]

2. Secondary Outcome: Overall Survival (OS) in the PDL-1 Positive Analysis Set
Description: OS is defined as the time from the date of randomization until the date of death due to any cause in the PD-L1 positive population, defined as vCPS ≥10%.
Time Frame: Through End-of-Trial Analysis data cutoff date of 28-Dec-2022 (up to approximately 5 years)
Population: The PD-L1 positive population included all randomized participants with tumor PD-L1 vCPS ≥10%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 80 | 62
Months | 10.2 [8.5 to 14.5] | 5.1 [3.8 to 8.2]

3. Secondary Outcome: Objective Response Rate (ORR) in the ITT Analysis Set
Description: ORR is defined as the percentage of participants who had complete response (CR) or partial response (PR) as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1;
Time Frame: Through End-of-Trial Analysis data cutoff date of 28-Dec-2022 (up to approximately 5 years)
Population: The ITT analysis set included all randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 256 | 256
Percentage of Participants | 20.3 [15.6 to 25.8] | 9.8 [6.4 to 14.1]

4. Secondary Outcome: Overall Response Rate (ORR) in the PD-L1 Positive Analysis Sets
Description: ORR is defined as the percentage of participants who had complete response (CR) or partial response (PR) as assessed by the investigator per RECIST v1.1;
Time Frame: Through End-of-Trial Analysis data cutoff date of 28-Dec-2022 (up to approximately 5 years)
Population: The PD-L1 positive population is defined as a visually-estimated combined positive score (vCPS) ≥10%
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 80 | 62
Percentage of Participants | 26.3 [17 to 37.3] | 11.3 [4.7 to 21.9]

5. Secondary Outcome: Progression-free Survival (PFS) in the ITT Analysis Set
Description: PFS is defined as the time from the date of randomization to the date of first documentation of disease progression assessed by the investigator per RECIST v1.1 or death, whichever occurs first; reported for the ITT analysis set
Time Frame: Through End-of-Trial Analysis data cutoff date of 28-Dec-2022 (up to approximately 5 years)
Population: The ITT analysis set included all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 256 | 256
Months | 1.6 [1.4 to 2.7] | 2.1 [1.5 to 2.7]

6. Secondary Outcome: Progression-free Survival (PFS) in the PDL-1 Positive Analysis Set
Description: PFS is defined as the time from the date of randomization to the date of first documentation of disease progression assessed by the investigator per RECIST v1.1 or death, whichever occurs first; reported for the PDL-1 Positive Analysis Set
Time Frame: Through End-of-Trial Analysis data cutoff date of 28-Dec-2022 (up to approximately 5 years)
Population: The PD-L1 positive population is defined as a visually-estimated combined positive score (vCPS) ≥10%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 80 | 62
Months | 2.7 [1.5 to 4.2] | 2.3 [1.4 to 3.0]

7. Secondary Outcome: Duration of Response (DOR) in the ITT Analysis Set
Description: DOR is defined as the time from the first determination of an objective response until the first documentation of progression as assessed by the investigator per RECIST v1.1, or death, whichever comes first
Time Frame: Through End-of-Trial Analysis data cutoff date of 28-Dec-2022 (up to approximately 5 years)
Population: The ITT analysis set included all randomized participants; only participants with an objective response (CR or PR) were included in this analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 52 | 25
Months | 7.1 [4.1 to 11.3] | 4.0 [2.1 to 8.2]

8. Secondary Outcome: Duration of Response (DOR) in the PDL-1 Positive Analysis Set.
Description: as for outcome 7
Time Frame: Through End-of-Trial Analysis data cutoff date of 28-Dec-2022 (up to approximately 5 years)
Population: The PD-L1 positive population is defined as a visually estimated combined positive score (vCPS) ≥10%; only participants with an objective response (CR or PR) were included in this analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 21 | 7
Months | 7.1 [2.9 to 13.2] | 5.7 [1.2 to NA] — Not estimable due to insufficient number of participants with events

9. Secondary Outcome: Health-Related Quality of Life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C-30) in the ITT Analysis Set
Description: Mean change from baseline in EORTC QLQ-C30 index score. The EORTC QLQ-C30 v3.0 is a questionnaire that assesses quality of life of cancer participants. It includes global health status and quality of life questions related to overall health in which participants respond based on a 7-point scale, where 1 is very poor and 7 is excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. A higher score indicates better health outcomes
Time Frame: Baseline to Cycle 6 (21 days per cycle)
Population: The ITT analysis set included all randomized participants; "Overall number of participants analyzed" refers to number of participants evaluable for this outcome measure and "Number analyzed" refers to participants evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 239 | 246
Score on a scale
  Baseline | 16.2 (12.28) | 18.3 (13.86)
  Change at Cycle 6: number analyzed (Participants) | 98 | 36
  Change at Cycle 6 | 0.2 (8.28) | 4.8 (9.38)

10. Secondary Outcome: HRQoL as Assessed by EORTC QLQ-C30 in the PDL-1 Positive Analysis Set
Description: as for outcome 9
Time Frame: Baseline to Cycle 6 (21 days per cycle)
Population: The PD-L1 positive population is defined as a visually estimated combined positive score (vCPS) ≥10%; "Overall number of participants analyzed" refers to number of participants evaluable for this outcome measure and "Number analyzed" refers to participants evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 77 | 59
Score on a scale
  Baseline | 16.8 (10.96) | 18.8 (12.02)
  Change at Cycle 6: number analyzed (Participants) | 39 | 9
  Change at Cycle 6 | 0.5 (7.39) | 0.5 (4.86)

11. Secondary Outcome: HRQoL as Assessed by EORTC QLQ-Oesophagus Cancer Module (EORTC QLQ-OES18) Reported in ITT Analysis Set
Description: Mean change from baseline in EORTC QLQ-OES18 index score. The EORTC QLQ-OES18 is a questionnaire that assesses overall symptoms in esophageal cancer participants. It includes questions related to overall health in which participants respond based on a 7-point scale, where 1 is very poor and 7 is excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. A higher score indicates better health outcomes.
Time Frame: Baseline to Cycle 6 (21 days per cycle)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 239 | 246
Score on a scale
  Baseline | 14.7 (11.81) | 16.3 (13.20)
  Change at Cycle 6 | -0.6 (8.63) | 3.0 (12.05)

12. Secondary Outcome: HRQoL as Assessed by EORTC QLQ-OES18) in the PDL-1 Positive Analysis Set.
Description: as for outcome 11
Time Frame: Baseline to Cycle 6 (21 days per cycle)
Population: The PD-L1 positive population is defined as a visually-estimated combined positive score (vCPS) ≥10%; "Overall number of participants analyzed" refers to number of participants evaluable for this outcome measure and "Number analyzed" refers to participants evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 76 | 59
Score on a scale
  Baseline | 16.5 (12.69) | 18.1 (12.21)
  Change at Cycle 6 | -0.9 (7.45) | -2.9 (5.16)

13. Secondary Outcome: HRQoL as Assessed by European Quality of Life 5-Dimensions 5-Level Questionnaire (EQ-5D-5L) in the ITT Analysis Set
Description: Mean change from baseline in EQ-5D-5L visual acuity score (VAS). The EQ-5D-5L measures health outcomes using a VAS to record a participant's self-rated health on a scale from 0 to 100, where 100 is 'the best health you can imagine' and 0 is 'the worst health you can imagine.' A higher score indicates better health outcomes.
Time Frame: Baseline to Cycle 6 (21 days per cycle)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 242 | 247
Score on a scale
  Baseline | 73.7 (17.05) | 72.5 (18.13)
  Change at Cycle 6 | -0.6 (14.81) | -5.9 (16.34)

14. Secondary Outcome: HRQoL as Assessed by EQ-5D-5L in the PD-L1 Positive Analysis Set
Description: as for outcome 13
Time Frame: Baseline to Cycle 6 (21 days per cycle)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 78 | 59
Score on a scale
  Baseline | 74.1 (14.84) | 70.5 (18.40)
  Change at Cycle 6 | -0.5 (17.59) | 4.4 (12.82)

15. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), which includes laboratory tests, physical exams, electrocardiogram results and vital signs
Time Frame: From the first dose date to 30 days after the last dose date; up to approximately 4 years and 11 months
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy
Number analyzed (Participants) | 255 | 240
Participants
  Number of participants with TEAEs | 245 | 236
  Number of participants with SAEs | 109 | 106

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events (AEs): up to approximately 4 years and 11 months
Description: All-cause mortality is reported for all randomized participants; Serious and other AEs include participants who received at least one dose of study drug.
  AEs are defined as events that had an onset date or a worsening in severity from baseline (pretreatment) on or after the first dose of study treatment up to 30 days following study treatment discontinuation or initiation of a new anticancer therapy, whichever occurred first.
Groups:
- Investigator Chosen Chemotherapy (ICC): Investigator choice of either paclitaxel 135-175 mg /m² on Day 1 IV every 21 days or 80-100 mg/m^2 on a weekly schedule; docetaxel 75 mg/m^2 IV on Day 1 every 21 days; or irinotecan 125 mg/m^2 IV on Days 1 and 8 every 21 days
Arm/Group | Tislelizumab | Investigator Chosen Chemotherapy (ICC)
All-Cause Mortality (participants affected / at risk) | 233/256 | 233/256
Serious Adverse Events (participants affected / at risk) | 109/255 | 106/240
Other Adverse Events (participants affected / at risk) | 232/255 | 231/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab (N=255) | Investigator Chosen Chemotherapy (ICC) (N=240)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 8 (9)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (7)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Autoimmune myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 13 (16) | 4 (5)
Gastric fistula (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 2 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (6)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 5 (6) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagomediastinal fistula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 3 (3) | 4 (5)
Malaise (General disorders) | 0 (0) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 3 (4) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Sudden death (General disorders) | 1 (1) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 19 (24) | 17 (18)
Pneumonia aspiration (Infections and infestations) | 3 (3) | 1 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (4) | 1 (1)
Septic shock (Infections and infestations) | 1 (2) | 4 (4)
Testicular abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 2 (3)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 10 (14)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 8 (11)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 6 (6)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (7) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to heart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (4)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (2)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Nephroangiosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab (N=255) | Investigator Chosen Chemotherapy (ICC) (N=240)
Anaemia (Blood and lymphatic system disorders) | 80 (139) | 109 (192)
Leukopenia (Blood and lymphatic system disorders) | 9 (19) | 29 (57)
Neutropenia (Blood and lymphatic system disorders) | 2 (11) | 30 (56)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7) | 10 (13)
Hyperthyroidism (Endocrine disorders) | 8 (8) | 1 (1)
Hypothyroidism (Endocrine disorders) | 30 (37) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 9 (10) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 17 (20) | 22 (27)
Abdominal pain upper (Gastrointestinal disorders) | 9 (12) | 16 (18)
Constipation (Gastrointestinal disorders) | 41 (46) | 45 (60)
Diarrhoea (Gastrointestinal disorders) | 32 (47) | 75 (134)
Dysphagia (Gastrointestinal disorders) | 22 (23) | 17 (22)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 (16) | 12 (13)
Nausea (Gastrointestinal disorders) | 37 (43) | 72 (123)
Stomatitis (Gastrointestinal disorders) | 9 (10) | 14 (21)
Vomiting (Gastrointestinal disorders) | 27 (33) | 48 (88)
Asthenia (General disorders) | 29 (41) | 36 (63)
Fatigue (General disorders) | 33 (43) | 42 (68)
Malaise (General disorders) | 16 (18) | 35 (54)
Oedema peripheral (General disorders) | 9 (12) | 11 (13)
Pyrexia (General disorders) | 40 (56) | 33 (42)
Nasopharyngitis (Infections and infestations) | 9 (14) | 6 (7)
Pneumonia (Infections and infestations) | 28 (31) | 14 (17)
Upper respiratory tract infection (Infections and infestations) | 8 (11) | 11 (11)
Alanine aminotransferase increased (Investigations) | 33 (49) | 19 (22)
Aspartate aminotransferase increased (Investigations) | 37 (55) | 11 (13)
Blood alkaline phosphatase increased (Investigations) | 17 (26) | 5 (10)
Blood bilirubin increased (Investigations) | 9 (16) | 6 (11)
Blood creatine phosphokinase MB increased (Investigations) | 11 (14) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 10 (15) | 0 (0)
C-reactive protein increased (Investigations) | 8 (8) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 14 (23) | 8 (10)
Lymphocyte count decreased (Investigations) | 12 (21) | 22 (36)
Neutrophil count decreased (Investigations) | 6 (19) | 88 (202)
Platelet count decreased (Investigations) | 14 (23) | 16 (20)
Weight decreased (Investigations) | 62 (101) | 45 (55)
White blood cell count decreased (Investigations) | 11 (25) | 95 (227)
White blood cell count increased (Investigations) | 12 (17) | 6 (8)
Decreased appetite (Metabolism and nutrition disorders) | 42 (53) | 80 (102)
Hyperglycaemia (Metabolism and nutrition disorders) | 17 (35) | 8 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (13) | 2 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 6 (13) | 11 (19)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 36 (51) | 30 (44)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (11) | 11 (17)
Hypochloraemia (Metabolism and nutrition disorders) | 6 (10) | 10 (13)
Hypoglycaemia (Metabolism and nutrition disorders) | 8 (11) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 22 (23) | 22 (42)
Hyponatraemia (Metabolism and nutrition disorders) | 31 (56) | 33 (45)
Hypoproteinaemia (Metabolism and nutrition disorders) | 13 (14) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (25) | 18 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (32) | 17 (27)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 14 (26)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (12) | 3 (4)
Dizziness (Nervous system disorders) | 11 (13) | 19 (26)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 23 (36)
Insomnia (Psychiatric disorders) | 21 (24) | 17 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 44 (56) | 28 (30)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (29) | 19 (23)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 5 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 18 (19)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 42 (46)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (34) | 11 (13)
Rash (Skin and subcutaneous tissue disorders) | 23 (31) | 10 (10)
Hypertension (Vascular disorders) | 13 (32) | 6 (15)
Hypotension (Vascular disorders) | 10 (14) | 6 (8)

LIMITATIONS AND CAVEATS:
The impact on treatment was considered very limited due to the small number of patients remaining on treatment, the short COVID-19 restriction period (in Asia), and limited restrictions for healthcare visits (in Europe/North America).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT03430843/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT03430843/SAP_001.pdf